CLINICAL TRIAL: NCT05763719
Title: Pathways to Improved Adolescent Mental Health Via an Economic and Gender Equality Intervention With Conflict Affected Families
Brief Title: Pathways to Improved Adolescent Mental Health in Conflict Affected Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: PAIDEK/Promotion de la Famille Paysanne (PFP) (Unknown); The Prevention Collaborative (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00368124; 5R01MH128913-02 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Mental Health Issue; Gender Equality
Keywords: Gender based violence; Economic empowerment; Couples intervention; Young adolescents
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rabbits for Resilience (RFR) + HIKA (Active Comparator): Households randomly selected for RFR + HIKA will consent to one adolescent (age 10-14 years) to participate in RFR, a youth led animal husbandry economic empowerment intervention, where each youth is provided training and mentorship on raising rabbits. Once the adolescent builds the rabbit cage, the adolescent receives a loan of 2 rabbits to raise and breed, once the rabbit produces offspring, the adolescent repays the rabbit loan with 2 rabbits, one to repay the loan and one to repay the interest on the loan. The original rabbits and the remaining offspring are then for the adolescents to continue to raise, breed, sell, or eat with mentorship from the RFR team and other family members. Parents (mother and father) will consent to complete a 22 week couple's curriculum to increase gender equality (e.g. shared decision making, improved communication and reduced partner violence). The curriculum is delivered for 3 hours weekly by trained facilitators with 12 couples per group.
  Interventions: Behavioral: Rabbits for Resilience (RFR) + HIKA
- Rabbits for Resilience (RFR) only (Active Comparator): Households randomly selected for RFR only will consent to one adolescent (age 10-14 years) to participate in RFR, a youth led animal husbandry economic empowerment intervention, where each youth is provided training and mentorship on raising rabbits. Once the adolescent builds the rabbit cage, the adolescent receives a loan of 2 rabbits to raise and breed, once the rabbit produces offspring, the adolescent repays the rabbit loan with 2 rabbits, one to repay the loan and one to repay the interest on the loan. The original rabbits and the remaining offspring are then for the adolescents to continue to raise, breed, sell, or eat with mentorship from the RFR team and other family members.
  Interventions: Behavioral: Rabbits for Resilience (RFR) only
- HIKA only (Active Comparator): Households randomly selected for HIKA, parents (mother and father) will consent to complete a 22 week couple's curriculum to increase gender equality (e.g. shared decision making, improved communication and reduced partner violence). The curriculum is delivered for 3 hours weekly by trained facilitators with 12 couples per group.
  Interventions: Behavioral: HIKA Healthy Relationship Program

INTERVENTIONS:
Behavioral: Rabbits for Resilience (RFR) + HIKA — Economic empowerment program using animal husbandry for young adolescents and healthy relationship program for parents/couples in same household
  Other Names: RFR + HIKA
  Arms: Rabbits for Resilience (RFR) + HIKA
Behavioral: Rabbits for Resilience (RFR) only — Economic empowerment program using animal husbandry with young adolescents
  Other Names: RFR only
  Arms: Rabbits for Resilience (RFR) only
Behavioral: HIKA Healthy Relationship Program — Healthy relationship program for parents/couples
  Other Names: HIKA only
  Arms: HIKA only

SUMMARY:
The study combined a youth-friendly economic empowerment program (Rabbits for Resilience (RFR) with a gender equality couple curriculum program (HIKA) to advance knowledge on the combined and synergistic impact of structural interventions and pathways with families for improved adolescent mental health in resource-poor communities. The investigators' multidisciplinary team will conduct a randomized controlled trial with three arms (RFR only, HIKA only, RFR + HIKA) with young adolescents ages 10-14 years and the adolescents' mothers and fathers living in 1080 rural households in 30 villages in two rural conflict-affected territories of South Kivu province of Eastern Democratic Republic of Congo (DRC)

DETAILED DESCRIPTION:
In the South Kivu province of the Democratic Republic of Congo (DRC), the setting for the study, families have experienced more than two decades of conflict and trauma, displacement and political instability resulting in extreme poverty with limited educational and economic opportunities. Child poverty and exposure to trauma is widespread and particularly concentrated in conflict-affected and hard-to-reach rural areas. According to UNICEF, 80% of DRC children have experienced at least two major deprivations (e.g., absences of food, housing, water, and medical care) in the children's lifetime. Childhood exposure to multiple adversities can lead to a lifetime of poor mental health. In the investigators' previous work in rural DRC, the investigators found parent's self-report of poor mental health and victimization or perpetration of intimate partner violence (IPV) had a significant negative impact on the parents' young adolescents' mental health and functioning, with different impacts for boys and girls. Specifically, mother's experience of IPV and symptoms of PTSD and depression had a stronger negative effect on adolescent girls in the household than on adolescent boys, including experienced stigma, externalizing behaviors, and school attendance. The underlying ideologies of male authority and of girls' and women's place being in the home has led to gender norms that restrict women and girl's mobility and opportunities. The impact of inequitable social norms on young adolescent mental health has had limited attention. Bolstering young peoples' mental health in the context of compounding childhood adversities and inequitable norms requires investments in families using locally designed and led multi-level interventions. The investigators' study will combine and examine the synergistic effect of two evidence-based interventions targeting young adolescents and the adolescents' mothers and fathers. Rabbits for Resilience (RFR) is a signature economic empowerment and mentorship program by the investigators' partner Congolese led non-governmental organization (NGO), Promotion de la Famille Paysanne (PFP). Young adolescents in RFR (with parent agreement) receive two rabbits and repay this asset loan with 2 offspring; these offspring are then provided as new assets to other youth in the same village, thus a sustainable program that also strengthens peer and family relationships. Adolescents and the adolescents' parents are mentored by RFR to continue to breed rabbits after repayment to sell or use to meet basic household needs (e.g. school fees, food), respond to economic shocks (e.g. illness) or opportunities (buy a goat). The investigators' randomized controlled trial demonstrated that adolescents in families active in RFR had improved mental health, enhanced food security and better school attendance.12 Harmful norms and behaviors, including a "husband's right to use violence to discipline his wife" have sustained inequalities and in the investigators' work influences who benefits most (boys or girls) from the RFR intervention. Therefore, RFR will be combined with HIKA meaning "to arrive". HIKA is an adapted 22 week group based, gender-equality curriculum delivered to couples/parents by trained local leaders. The HIKA program strengthens family relations through knowledge and skills building in communication, power sharing, parenting, and conflict management. Couples participating in the program in Rwanda reported less physical and/or sexual violence victimization and perpetration over a 24-month period. Additional benefits included reductions in acceptability of wife beating, conflict with partner, corporal punishment, depression and improved communication, self-efficacy and self-rated health. Combining a youth-friendly economic empowerment program with a gender equality program with parents of these young adolescents will advance knowledge on the combined and synergistic impact of structural interventions and pathways for improved adolescent mental health. The investigators' multidisciplinary team will conduct a clustered randomized controlled trial with three arms (RFR only, HIKA only, RFR + HIKA) with young adolescents ages 10-14 years and the adolescents' parents living in 1080 rural households in 30 villages in two rural conflict-affected territories of South Kivu province of Eastern DRC.

1. Examine the combined and synergetic effect of RFR and HIKA on young adolescent mental health. Hypothesis 1. Adolescents in RFR + HIKA households will report greater improvement in mental health compared to adolescents in RFR only and HIKA only households in rural conflict affected villages.
2. Examine the pathways through which RFR and HIKA improves adolescent mental health.

   * Hypothesis 2a. Adolescents in the RFR + HIKA and RFR households will report greater improvement in mental health via pathway of improved self-efficacy, school attendance, food security and peer relationships compared to adolescents in HIKA only households in rural conflict-affected villages.
   * Hypothesis 2b. Adolescents in RFR + HIKA and HIKA only households will report greater improvement in mental health via the pathway of improved parental (mother and father) relationship quality and power sharing, reduced exposure to IPV/corporal punishment, improved parental mental health and support of gender equitable norms compared to adolescents in RFR only households in rural conflict affected villages.
3. Examine if the pathways by which RFR and HIKA improve adolescent mental health differ by sex.

ELIGIBILITY:
Inclusion Criteria:

* Resident in household located in one of 30 villages in 2 territories in South Kivu province in Eastern DRC
* One adolescent (boy or girl) age 10-14 years living in household
* Mother and father (parents or guardians) of eligible adolescent living in same household
* Family plans to remain residents in the village for next 18 months
* Parents/guardians (mother and father) consent to participate in 22 week couple curriculum
* Adolescent consents to participate in animal husbandry economic empowerment program

Exclusion Criteria:

* Household members planning to move or leave the study village in next 18 months
* Household does not have a boy or girl age 10-14 years living in it
* Mother and/or father (parents or guardians) are not living in the household
* Parents/guardian do not consent to participate in 22 week couple curriculum
* Adolescent does not consent to participate in the animal husbandry economic empowerment program

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3024 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in adolescent Mental Health as assessed by Kidscreen | Baseline, 3, 6 and 12 months
  Kidscreen Psychological Well-Being is on a 1 to 5 scale with higher scores representing better psychological well-being

SECONDARY OUTCOMES:
Change in Adolescent Economic Empowerment assessed by 5 economic skills items | Baseline, 3, 6, and 12 months
  is on a 1 to 5 scale with higher scores representing greater economic empowerment
Change in Adolescent Food Security as assessed by the Household Food Insecurity Access Scale | Baseline, 3, 6 and 12 months
  Household Food Insecurity Access Scale is on a 1 to 4 with higher scores representing greater food insecurity
Change in Parent Relationship and Home Life as assessed on Kidscreen | Baseline, 3, 6 and 12 months
  Kidscreen Psychological Well-Being is on a 1 to 5 scale with higher scores representing better relationships

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Glass, PhD, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins University School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, behavioral and clinical data will be collected using two (Adult and Adolescent) preprogrammed surveys using the secure Redcap platform based and managed by Johns Hopkins University. A planned 1080 male and female adolescents ages 10-14 will provide data across 4 time points (baseline, 3, 6 and 12 months post baseline). Demographic, behavioral and clinical data will be collected from 1080 couples/parents (1080 male/fathers and 1080 female/mothers) across 4 time points (baseline, 3, 6, and 12 months). Therefore, demographic, behavioral and clinical data will be collected from a total of 3,240 adults and adolescents over 12 months. All data will be de-identified prior to receipt in the repository, but the information needed to generate a global unique identifier for National Institute of Mental Health (NIMH) Data Archiver (NDA) will be collected for each study participant.
Supporting Information: Study Protocol
Time Frame: The baseline data will be deposited in the NDA by July 1, 2023 (approximately 4 months after data collection). Thereafter, scientific data will be deposited on January 1 and July 1 (standard NDA dates). NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.
Access Criteria: Data will be findable for the research community through the NDA Collection established for this study. For all publications, an NDA study will be created. Each of those studies is assigned a digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication.
  As required by NDA, studies will also be created that contain the data used for every publication. Those studies will be shared when the pre-print is available. NDA studies have digital object identifiers (DOI) to aid in finding. The investigators will include that DOI in relevant publications.